CLINICAL TRIAL: NCT01898390
Title: An Open Label Study to Assess the Safety and Efficacy of Neural Allo-Transplantation With Fetal Ventral Mesencephalic Tissue in Patients With Parkinson's Disease
Brief Title: TRANSEURO Open Label Transplant Study in Parkinson's Disease
Acronym: TRANSEURO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Lund University (Other); Cardiff University (Other); Imperial College London (Other); University College, London (Other); University Hospital Freiburg (Other); Life Science Governance Institute (Unknown); Assistance Publique - Hôpitaux de Paris (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Life Technologies Ltd, part of Thermo Fisher Scientific (Unknown); Inomed (Unknown); Cambridge Cognition Ltd (Industry); Skane University Hospital (Other); Imanova Limited (Unknown)
Responsible Party: Principal Investigator, Prof Roger Barker, Professor, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANSEURO; FP7-242003 (Other Grant/Funding Number: European Community Seventh Framework Programme)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Allo-Transplantation; Fetal Ventral Mesencephalic Tissue
MeSH Terms: conditions — Parkinson Disease | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transplant (Experimental): Neural Allo-Transplantation with Fetal Ventral Mesencephalic Tissue
  Interventions: Procedure: Transplant
- Control (No Intervention): comparison group of controls, will receive the same observational and scanning assessments but will not receive any surgical procedures

INTERVENTIONS:
Procedure: Transplant — Bilateral Neural Allo-Transplantation with Fetal Ventral Mesencephalic Tissue
  Arms: Transplant

SUMMARY:
The Transeuro Transplant study is a trial which will involve grafting foetal tissue into the brain of patients with Parkinson's disease, who are already been followed in the observational study. The tissue inserted in the brain is to help replace and rebuild lost dopamine from the brain due to Parkinson's disease.

Update April 2019:

A total of 11 PD patients were grafted in Cambridge, UK and Lund, Sweden. No further surgeries are planned. The final patient will complete the study's clinical endpoint (36 months post-graft) in 2021. We continue to assess these patients bi-annually alongside a control group which did not receive any intervention.

DETAILED DESCRIPTION:
Clinical trials of cell therapy in PD patients were first performed in Lund in the late 1980s, followed by a number of similar, small trials in other European and North American centres. These initial studies performed on small groups of advanced PD patients were all open label but firmly established safety of the procedure. The results obtained in these trials have shown that the grafted dopaminergic [DA] neurons can survive and function long-term, over more than 10 years, and that some patients have shown clear clinical benefits, especially with respect to their bradykinesia and rigidity, with reductions in L-dopa requirements. Using functional imaging it has also been shown that the grafted DA neurons can restore striatal DA release and provide a sustained re-activation of motor cortical areas, i.e. key areas that were underactive prior to grafting.

Post-mortem studies have shown excellent long-term survival of the grafted DA neurons, notwithstanding the observation that some of the long-term surviving transplants (at 12-15 years after grafting) have now been shown to contain signs of PD-related pathologies, i.e. neuronal Lewy-bodies and alpha-synuclein positive inclusions in the grafts. However, such changes have been observed only in some and not in all patients and when seen the extent of the pathology is limited to a small number of the grafted DA cells and the clinical consequence, if any, not known.

However, the outcomes of two NIH sponsored double blind placebo controlled trials, which published their main findings in 2001 and 2003, have raised major concerns. In both these trials the grafted patients did not show any significant improvement overall compared to sham-operated controls at 1 and 2 years post grafting. Furthermore, a significant number of patients in both trials developed GIDs, which in some cases were so severe that further neurosurgery was needed to remedy the situation.

The reasons for the variable, and overall poor, outcome in these trials, including the generation of GIDs, have been the subject of much debate but have recently centred on three key elements, with an additional possible fourth element:

* The selection of patients in terms of clinical phenotype, disease stage and pattern of striatal dopaminergic denervation at the time of grafting;
* The differences in immunosuppressive regimes and the risk that incomplete immunosuppression in combination with the use of solid graft methods may lead to the development of detrimental immune/inflammatory reactions at the graft site with compromise of the grafted dopamine cell function;
* The mode of engraftment and differences in graft cell survival, and the risk for inhomogeneous delivery of dopaminergic neurons and the generation of potentially dyskinesia-inducing "patchy" innervations in the host striatum;
* A final possible element is the composition of the grafted tissue and the ratio of serotoninergic to dopaminergic neurons within the graft. There is emerging evidence that serotoninergic neurons can release dopamine in a relatively unregulated fashion given they lack transporters for it, and as such may use L-dopa as a false transmitter which may not only underlie the development of L-dopa induced dyskinesia's but may also contribute to GIDs.

Failure of the NIH trials to demonstrate any overall clinical benefits in the grafted patients, and the unexpected and worrisome development of GIDs in a significant number of patients in these trials has represented a major hurdle for the future development of cell based therapies for PD and it is in this and related areas that this project seeks to move the field forward and go beyond the current state of the art for this treatment approach.

This project has gathered together all the available expertise in this area to resolve or reduce the risk of the previous complications seen with VM transplants in patients with PD. We will conduct a new round of clinical trials, involving a step-by-step optimisation of all technical aspects of the grafting procedure and patient selection and assessment, in order to improve clinical efficiency and consistency, in the absence of troublesome dyskinesia's.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet ALL of the following criteria to be considered for the enrolment into this study:

  * PD as defined using Queen's Square Brain Bank criteria.
  * Disease duration ≥ 2 years and ≤ 13 years.
  * Aged ≥ 30 years and ≤ 68 years at the time of grafting.
  * Hoehn & Yahr stage 2.5 or better when 'on'.
  * On standard anti PD medication without significant LIDs defined as a score of >2 on the AIMS dyskinesia rating scale, in any body part.
  * Patients must be right handed.

Exclusion Criteria:

* Any of the following will exclude patients from being enrolled in the study:

  * Atypical or secondary parkinsonism including F-DOPA PET patterns consistent with this.
  * Clinically significant response to Levodopa (as evaluated by the clinician) and/or apomorphine challenge.
  * Mini-Mental State Examination (MMSE) score of less than 26.
  * Unable to do normal copying of interlocking pentagons and semantic fluency score for naming animals of less than 20 over 90 seconds as these have recently been associated with the earlier onset of dementia in PD.
  * Ongoing major medical or psychiatric disorder including depression and psychosis.
  * Other concomitant treatment with neuroleptics (inc. Atypical neuroleptics) and cholinesterase inhibitors.
  * Significant drug induced dyskinesia defined as a score of >2 on the AIMS dyskinesia rating scale, in any body part.
  * Previous neurosurgery, cell therapy or organ transplantation.
  * Unable to be imaged using MRI.
  * Any contraindication to immunosuppression therapy.
  * Patients on anticoagulants
  * Patients who are left handed

Ages: 30 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-05; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in UPDRS score | 36 months post transplantation
  The change in motor Unified Parkinson's Disease Rating Scale (UPDRS)in a defined "OFF" state at 36 months post transplantation. "OFF" being defined as receiving no dopamine (DA) therapy for 12 hours prior to assessment or longer in the case of long acting dopamine agonists (e.g. Ropinirole slow release).

SECONDARY OUTCOMES:
Change in timed motor tasks | 36 months post transplantation
  Change in timed motor tasks at 36 months post transplantation
Number of dyskinesias at 36 months | 36 months post transplantation
  The number of patients with dyskinesias (including L-dopa and graft induced dyskinesias) at 36 months post transplantation
L-dopa equivalent medication at 36 months | 36 months post transplantation
  L-dopa equivalent medication doses at 36 months post transplantation.
L-dopa therapy at 36 months | 36 months post transplant
  Number of patients on L-dopa therapy at 36 months post transplantation.
Off time medication at 36 months | 36 months post transplantation
  The amount of 'off' time 36 months post transplantation
Quality of life change at 36 months | 36 months post transplantation
  Quality of life (change) 36 months post transplantation
F-DOPA PET changes | 36 months post transplantation
  Changes in F-DOPA PET in transplanted patients 36 months post transplantation

OTHER OUTCOMES:
AE/SAE's | 0-36 months post treatment
  The number of adverse events and serious adverse events associated with the neural transplant
Laboratory Parameters | 0-36 months post treatment
  Any reported changes in haematology, biochemistry or urinalysis measures outside the normal range
Other Safety parameters | 0-36 months post treatment
  Vital signs, Physical Exam - new abnormalities will be recorded as an adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Roger Barker, Prof, Principal Investigator — Department of Clinical Neurosciences, University of Cambridge